CLINICAL TRIAL: NCT00816309
Title: Is Regular Chest Physiotherapy an Effective Treatment in Severe, Non Cystic Fibrosis Bronchiectasis?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Dr Adam Hill, Consultant Respiratory Physician, NHS Lothian, NHS Lothian
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AH003
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2010-07

CONDITIONS: Bronchiectasis
Keywords: physiotherapy; bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acapella Physiotherapy (Experimental): Physiotherapy with acapella versus no physiotherapy
  Interventions: Device: Acapella Physiotherapy
- No physiotherapy (No Intervention): Physiotherapy with acapella versus no physiotherapy

INTERVENTIONS:
Device: Acapella Physiotherapy — twice daily- around 20 minutes
  Arms: Acapella Physiotherapy

SUMMARY:
Bronchiectasis is a chronic chest condition which causes a persistent cough and frequent chest infections. One of the main forms of treatment is chest physiotherapy. Physiotherapy is thought to improve cough and help clear the airways of sticky sputum. Traditionally, physiotherapy techniques can be awkward, but recently a new device (a simple mouthpiece, called the Acapella device) has been developed to make physiotherapy practise easier. This study aims to assess how helpful regular physiotherapy using a new mouthpiece is in patients with severe bronchiectasis.

DETAILED DESCRIPTION:
Study being carried out in the Department of Respiratory Medicine, Royal Infirmary of Edinburgh.

The study is entitled "Is regular chest physiotherapy an effective treatment in severe, non cystic fibrosis bronchiectasis?" This is a small randomised controlled pilot crossover study assessing the efficacy of regular chest physiotherapy using an Acapella mouthpiece in severe non cystic fibrosis bronchiectasis. 10 patients will be randomised to receive full instruction in use of the Acapella device (twice daily therapy) and ten patients will continue with their standard treatment regimen. The study will be conducted over seven months.

At the beginning we will randomly allocate them to receive either the current standard treatment regimen for bronchiectasis or to receive instruction in the use of the Acapella physiotherapy device for the first 3 months.

After these 3 months all will receive the current standard treatment regimen for 1 month.

Following this, those that received current standard treatment will receive Acapella physiotherapy device for 3 months and those that received Acapella physiotherapy device will stop this and receive current standard treatment for 3 months.

All participants will be reviewed on 6 occasions (start of study and then at months 1, 2, 3, 4 and 6). At each review, sputum samples will be collected, routine bloods, spirometry and exercise testing performed and health related quality of life questionnaires be completed.

At the end of the study should patients have felt benefit with the physiotherapy with the Acapella device, they should continue using it regularly on a twice-daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Moderate and Severe Bronchiectasis
* No regular chest physiotherapy

Exclusion Criteria:

* Moderate or Severe COPD

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
24 hour sputum volume and assessment of cough severity (Leicester Cough Questionnaire) | 3 months

SECONDARY OUTCOMES:
spirometry (FEV1, FVC, FEF 25-75), incremental shuttle test, St George's Respiratory Questionnaire and Nottingham Health Profile NHP-2, quantitative bacteriology. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Hill, MBChB MD, Principal Investigator — NHS Lothian
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Murray MP, Pentland JL, Hill AT. A randomised crossover trial of chest physiotherapy in non-cystic fibrosis bronchiectasis. Eur Respir J. 2009 Nov;34(5):1086-92. doi: 10.1183/09031936.00055509. Epub 2009 Jun 18. PMID 19541717